CLINICAL TRIAL: NCT02504697
Title: Detection of Early Lung Cancer Among Military Personnel Study 2 (DECAMP-2): Screening of Patients With Early Stage Lung Cancer or at High Risk for Developing Lung Cancer
Brief Title: DECAMP-2: Screening of Patients With Early Stage Lung Cancer or at High Risk for Developing Lung Cancer
Acronym: DECAMP-2
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Other Study IDs: H-32479
Record Dates: First submitted 2014-05-27; First posted 2015-07-22 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Sputum, Nasal brushing, Buccal scraping, Bronchial Biopsy, Bronchial brushing, lung tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Longitudinal Cohort: For this longitudinal screening cohort, we will enroll 800 participants who currently or historically smoked and who have a 10 year Bach risk model of lung cancer > 2.5% (5). We will include participants 50 to 79 years old, with ≥10 cigarettes/day for current smokers, or ≥20 pack years for former smoker who quit 20 years ago or less. In order to further enrich for lung cancer risk, participants also will have COPD/emphysema or at least one first-degree relative with a diagnosis of lung cancer. We will exclude patients previously diagnosed with lung cancer. These patients will be followed for a total of 4 years with annual follow-up visits. Biosamples from airway and blood and images will be collected.
  Interventions: Other: Biosamples from airway and blood

INTERVENTIONS:
Other: Biosamples from airway and blood — Identify biomarkers in biosamples from airway and blood for the preclinical detection of lung cancer.

SUMMARY:
The goal of this project is to improve lung cancer screening in high-risk individuals by identifying biomarkers of preclinical disease and disease risk that are measured in minimally invasive and non-invasive biospecimens. Existing biomarkers for lung cancer diagnosis as well as new biomarkers discovered specifically in this clinical setting will be examined. Biomarkers that identify individuals at highest risk for being diagnosed with lung cancer prior to the appearance of concerning symptoms could increase the utility of lung cancer surveillance and the efficiency of lung cancer chemoprevention clinical trials. Achieving these goals would improve the detection and treatment of early stage and incipient lung cancer, while restricting the risk of these procedures to those individuals who currently exhibit the early molecular warning signs of impending disease.

DETAILED DESCRIPTION:
The Detection of Early lung Cancer Among Military Personnel (DECAMP) consortium is a multidisciplinary and translational research program that includes 7 Veterans Administration Hospitals (VAH), the 4 designated Military Treatment Facilities (MTF) and 4 academic hospitals as clinical study sites, several molecular biomarker laboratories, along with Biostatics, Bioinformatics, Pathology and Biorepository cores. The DECAMP Coordinating Center will facilitate rapid selection, design and execution of clinical studies within this multi-institutional consortium. The ACRIN 4704 study will recruit one cohort to achieve the aims of this study: a longitudinal screening cohort.

ELIGIBILITY:
Inclusion Criteria for longitudinal screening cohort

* Ages 50 to 79 years;
* Smoking status: Current or former smoker (≥10 cigarettes/day for current smokers, or ≥20 pack years for former smoker who quit 20 years ago or less)
* History of Chronic Obstructive Pulmonary Disease (COPD), emphysema, or at least one first-degree relative with a diagnosis of lung cancer;
* Willing to undergo fiberoptic bronchoscopy;
* Able to tolerate all biospecimen collection as required by protocol;
* Able to comply with standard-of-care follow-up visits, including clinical exams, diagnostic work-ups, and imaging for a maximum of four years or until diagnosis of lung cancer;
* Able to fill out Patient Lung History questionnaire;
* Willing and able to provide a written informed consent.

Exclusion Criteria

* Diagnosis of lung cancer prior to the current assessment (that is, patients are eligible if first lung cancer diagnosis has been recently confirmed by bronchoscopic biopsy and is leading to resection surgery, but not if this is not a first diagnosis);
* Contraindications to nasal brushing or fiberoptic bronchoscopy, including: ulcerative nasal disease, hemodynamic instability, severe obstructive airway disease (i.e., disease severity does not allow for bronchoscopic procedures), unstable cardiac or pulmonary disease, as well as other comorbidities leading to inability to protect airway, or altered level of consciousness;
* Allergies to any local anesthetic that may be used to obtain biosamples in the study;
* Weight greater than that allowable by the CT scanner.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Military personnel
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer | Four years

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Billatos, MD, Principal Investigator — Boston University; Denise Aberle, MD, Principal Investigator — University of California, Los Angeles
Locations (15):
- United States (15):
  - Regents of the University of California LA (Los Angeles VA Healthcare System), Los Angeles, California
  - University of California Los Angeles Medical Center, Los Angeles, California
  - Naval Medical Center San Diego, San Diego, California
  - Denver Research Institute, Denver, Colorado
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Boston VA Research Institute, Inc, Boston, Massachusetts
  - Health Research Inc. Roswell Park Division, Buffalo, New York
  - Trustees of University of Pennsylvania (Philadelphia VA Medical Center), Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Veterans Research Foundation of Pittsburgh, Pittsburgh, Pennsylvania
  - Middle Tennessee Research Institute (Vanderbilt University), Nashville, Tennessee
  - Dallas VA Research Corporation, Dallas, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Billatos E, Ash SY, Duan F, Xu K, Romanoff J, Marques H, Moses E, Han MK, Regan EA, Bowler RP, Mason SE, Doyle TJ, San Jose Estepar R, Rosas IO, Ross JC, Xiao X, Liu H, Liu G, Sukumar G, Wilkerson M, Dalgard C, Stevenson C, Whitney D, Aberle D, Spira A, San Jose Estepar R, Lenburg ME, Washko GR; DECAMP and COPDGene Investigators. Distinguishing Smoking-Related Lung Disease Phenotypes Via Imaging and Molecular Features. Chest. 2021 Feb;159(2):549-563. doi: 10.1016/j.chest.2020.08.2115. Epub 2020 Sep 16. PMID 32946850
- [Derived] Billatos E, Duan F, Moses E, Marques H, Mahon I, Dymond L, Apgar C, Aberle D, Washko G, Spira A; DECAMP investigators. Detection of early lung cancer among military personnel (DECAMP) consortium: study protocols. BMC Pulm Med. 2019 Mar 7;19(1):59. doi: 10.1186/s12890-019-0825-7. PMID 30845938